CLINICAL TRIAL: NCT05077709
Title: A Phase II Multi-Arm (Basket) Trial Investigating the Safety and Efficacy of IO102-IO103 in Combination With Pembrolizumab, as First-Line Treatment for Patients With Metastatic NSCLC, SCCHN, or Metastatic mUBC
Brief Title: IO102-IO103 in Combination With Pembrolizumab as First-line Treatment for Patients With Metastatic NSCLC, SCCHN, or mUBC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IO Biotech (Industry)
Collaborators: Theradex (Industry); Almac (Industry); NeoGenomics (Unknown); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOB-022; KEYNOTE-D38 (Other: Merck)
Record Dates: First submitted 2021-09-09; First posted 2021-10-14 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer Non Small Cell; Head and Neck Squamous Cell Carcinoma; Urothelial Carcinoma Bladder
Keywords: NSCLC; SCCHN; mUCB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: All participants receive IO102-IO103 for three different indications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (NSCLC) (Experimental): NSCLC patients (metastatic stage IV) treated with IO102-IO103 SC Q3W in combination with pembrolizumab IV 200mg Q3W
  Interventions: Drug: IO102-IO103 in combination with pembrolizumab
- Arm B (SCCHN) (Experimental): SCCHN patients (metastatic stage IV) treated with IO102-IO103 SC Q3W in combination with pembrolizumab IV 200mg Q3W
  Interventions: Drug: IO102-IO103 in combination with pembrolizumab
- Arm C (mUBC) (Experimental): mUBC patients (metastatic stage IV) treated with IO102-IO103 SC Q3W in combination with pembrolizumab IV 200mg Q3W
  Interventions: Drug: IO102-IO103 in combination with pembrolizumab

INTERVENTIONS:
Drug: IO102-IO103 in combination with pembrolizumab — The experimental drug IO102-IO103 is for SC injection and consist of IDO and PD-L1 peptides

SUMMARY:
A Phase II Multi-Arm (basket) Trial Investigating the Safety and Efficacy of IO102-IO103 in Combination with pembrolizumab, as First-line Treatment for Patients with Metastatic Non-Small Cell Lung Cancer (NSCLC), Squamous Cell Carcinoma of Head or Neck (SCCHN), or Metastatic Urothelial Bladder Cancer (mUBC)

DETAILED DESCRIPTION:
Naturally occurring IDO/PD-L1 specific T-cells recognize MHC-bound IDO/PD-L1 peptides, and are able to eliminate IDO expressing or PD-L1 expressing immune regulatory cells and cancer cells. Activation of IDO or PD-L1 specific T-cells through vaccination with the IDO and PD-L1 peptides (IO102-IO103) will boost natural killing of cancer cells and counteract immune regulatory mechanisms in the tumor microenvironment. Thus, IDO/PD-L1 specific T-cells may both directly support anti-cancer immunity by killing target T-cells but also indirectly by releasing pro-inflammatory cytokines in the microenvironment to boost additional anti-cancer immunity.

This is a non comparative, open label, unblinded, multi-arm (basket) trial of IO102-IO103 in combination with pembrolizumab in three indications: NSCLC, SCCHN or mUBC. The primary objective of the trial is to investigate the efficacy of IO102-IO103 in combination with pembrolizumab in the frontline treatment in each of the different metastatic solid tumour indications with the intent to expand a specific arm if a clinically meaningful signal is observed based on primary endpoint (dual target of either ORR or PFS by investigator assessment according to RECIST v.1.1).

Approximately 90 patients will be enrolled and treated; approximately 30 patients in each arm. All eligible patients will receive treatment for up to 2 years with IO102-IO103 (IO102 85μg and IO103 185μg) SC Q3W in combination with pembrolizumab IV 200mg Q3W.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed:

   Metastatic NSCLC (Arm A), who have not received prior systemic treatment for their metastatic disease and who have:

   • no known sensitizing EGFR or ALK mutations.

   or

   Metastatic SCCHN (Arm B) with no prior therapy and who have:

   • Histologically- or cytologically-confirmed recurrent or metastatic SCCHN considered incurable by local therapies. Tumors of nasopharyngeal origin (any histology) are excluded

   • Documented results of HPV status for oropharyngeal cancer.

   or

   Metastatic UBC (Arm C) with no prior therapy and not eligible for any cisplatin therapy:

   • Advanced/unresectable (inoperable) or metastatic urothelial cancer of the renal pelvis, ureter, bladder or urethra (transitional cell and mixed transitional/non transitional cell histologies permitted but transitional cell histology must be the dominant histology)

   All solitary metastases must be biopsied to confirm diagnosis of metastases from primary indication
2. PD-L1 tumor expression or PD-L1 CPS (as confirmed prior to enrolment using the DAKO 22C3 assay, using local/central services):

   • Arm A (NSCLC): PD-L1 TPS ≥ 50%

   • Arm B (SCCHN): PD-L1 CPS ≥ 20; HPV +/-

   • Arm C (mUBC): PD-L1 CPS ≥ 10
3. A male participant able to father a child must agree to use contraception starting with the screening visit and through 120 days after last dose of pembrolizumab or 180 days after last dose of treatment with IO102-IO103.
4. A female participant is eligible to participate if she is not pregnant not breastfeeding, and at least one of the following conditions applies:

   • Not a woman of childbearing potential (WOCBP)

   • A WOCBP who agrees to follow contraceptive guidance starting with the screening visit and through 120 days after last dose of pembrolizumab or 180 days after last dose of chemotherapy.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial in accordance with ICH-GCP and local legislation prior to admission to the trial.
6. At least 18 years of age on day of signing informed consent
7. Have measurable disease per RECIST 1.1 as assessed by local site investigator/radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have provided a blood sample and archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded tissue blocks are preferred to slides.
9. Have an ECOG performance status of 0 to 1.
10. If participant received major surgery, they must have recovered adequately from the adverse events and/or complications from the intervention prior to starting trial treatment.
11. Have adequate organ function as defined in the protocol. Specimens must be collected within 10 days prior to the start of trial treatment.Have adequate organ function as defined below. Specimens must be collected within 10 days prior to the start of trial treatment.

    Adequate organ function as defined by:
    * Haematology:

    Absolute neutrophil count ≥ 1500/µL or ≥ 1.5 x 109/L Platelets ≥ 100,000/µL or ≥ 100 x 109/L Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L • Renal: Creatinine ≤ 1.5 x ULN, or Measured or calculated creatinine clearance (CrCl) ≥ 60 mL/min for patients with creatinine levels > 1.5 x institutional ULN; GFR can also be used in place of creatinine or CrCl • Hepatic: Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels ≤3 x ULN AST and ALT ≤ 2.5 x ULN (≤ 5xULN for patients with liver metastases) Alkaline Phosphatase ≤ 2.5 x ULN

    • Endocrine: Thyroid stimulating hormone (TSH) within normal limits, or Total T3 is within normal limits, or Free T3 and free T4 are within the normal limits
    * Coagulation:

    International normalised ratio, PT or aPTT ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

    Exclusion Criteria:

<!-- -->

1. A WOCBP who has a positive urine pregnancy test (e.g., within 72 hours) prior to treatment. If at any time, a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137) other than for adjuvant or neoadjuvant treatment AND was discontinued from that treatment due to a Grade 3 or higher immune-related AE (irAE).
3. Has received prior systemic anti-cancer therapy in the first line setting for the participant's metastatic disease (treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 6 months prior to diagnosis of metastatic disease).
4. Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy are eligible.
5. Has received prior radiotherapy to the lung >30 Gy within 6 months of start of trial treatment and have recovered from all radiation-related adverse events, not have require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
6. Have a life expectancy of < 3 months and/or rapidly progressing disease.
7. Have received a live or live attenuated vaccine within 30 days prior to the first dose of trial treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
8. Participation in or has participated in a trial of an investigational agent within 30 days prior to study entry or has used an investigational device within 6 months prior to the first dose of trial treatment. Note: Participants who have entered the follow-up phase of an investigational trial may participate as long as it has been 6 months after the last dose of the previous investigational agent.
9. Has a diagnosis of immunodeficiency10. Received any of the following medications or procedures within 2 weeks prior to time of treatment initiation: Systemic or topical corticosteroids at immunosuppressive doses > 10 mg/day of hydrocortisone or > 5mg/day of prednisone equivalent.
10. Has a known additional malignancy that is progressing or has required active treatment within the past 2 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
11. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during trial screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of trial treatment.
12. Has severe hypersensitivity (≥Grade 3) to IO102 or IO103, pembrolizumab and/or any of their excipients.
13. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
14. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
15. Has an active infection requiring systemic therapy.
16. Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority.
17. Known adrenal insufficiency function (that is basal cortisol level < 140nmol/L or < 5 μg/dL).
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV) (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection.
19. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the trial.
21. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 180 days after last dose of trial treatment.
22. Has had an allogenic tissue/solid organ transplant.
23. Has progressive disease (PD) within six months of completion of curatively intended systemic treatment for locoregionally advanced SCCHN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
ORR or PFS | 6 months
  Target ORR according to RECIST v1.1 or PFS Rate at 6 months as per investigator assessments.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  PFS is defined as the time from first treatment with IMP to the first documented disease progression (based on disease evaluation done locally for all patients in accordance with RECIST v.1.1) or death from any cause. If a patient is not known to have progressed or died then they will be censored at the date of the last disease assessment. If a patient progresses after they have 2 or more missed disease assessment visits then they will be censored at the date of the last non missing disease assessment.
Duration of Response (DoR) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  DoR will be measured from the date of first observed objective response until disease progression or death (whichever is earlier). Date of progression and censoring will be handled in the same way as for PFS (evaluation done locally for all patients in accordance with RECIST v.1.1). The time of the initial response will be defined as the latest of the dates contributing towards the first visit response of PR or CR. If a patient does not progress following a response, then their duration of response will use the PFS censoring time.
Complete Response Rate (CRR) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  CRR is defined as the number (%) of patients with a visit response of CR. Evaluation of response will be done locally for all patients in accordance with RECIST v.1.1.
Disease Control Rate (DCR) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  DCR is defined as the number (%) of patients with a visit response of PR or CR or SD. Evaluation of response will be done locally for all patients in accordance with RECIST v.1.1.
Overall Survival (OS) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  Overall survival is defined as the time from first dose of IMP until death from any cause. Patients not known to have died will be censored at the date last known to be alive. After disease progression, all patients are expected to be followed every 12 weeks to confirm their survival status. These follow-up visits/contacts continue until the last planned overall survival analysis.
Time to Response (TTR) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  In the subset of responding patients, TTR is defined as the time from first dose of IMP until the date of the first observed partial or complete response. Evaluation of response will be done locally for all patients in accordance with RECIST v.1.1.
Safety reporting | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  AE/SAE collection

OTHER OUTCOMES:
Exploratory Endpoint: Biomarkers | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  Biomarkers will be assessed and correlated both to the clinical response (after treatment) and the induced immunological response
Exploratory Endpoint: Progression Free Survival according to iRECIST (iPFS) | Every 9 weeks during the first year of treatment and then every 12 weeks for the second year of treatment
  PFS is defined as the time from first treatment with IMP to the first documented disease progression (based on iRECIST) or death from any cause. Per iRECIST disease progression should be confirmed by the site 4 to 8 weeks after site-assessed first radiologic evidence of PD (iUPD). The event date used for calculation for progression free survival should be the first date progression criteria is met (iUPD) providing that progression is confirmed at the next assessment.If a patient is not known to have progressed or died then they will be censored at the date of the last disease assessment. If a patient progresses after they have 2 or more missed disease assessment visits then they will be censored at the date of the last non missing disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Riess, MD, MSc, Principal Investigator — Division of Hematology/Oncology, UC Davis Comprehensive Cancer Center
Locations (21):
- United States (9):
  - City of Hope, Duarte, California
  - UC Davis Cancer Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Montefiore Medical Center, The Bronx, New York
  - University of Toledo Medical Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Cancer Specialists, Fairfax, Virginia
- Spain (10):
  - Hospital Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia (ICO) Badalona (Catalan Institute of Oncology), Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza
- United Kingdom (2):
  - Velindre Cancer Center, Cardiff
  - Guys and St Thomas Hospital, London